CLINICAL TRIAL: NCT06583239
Title: Developing and Evaluating a Hub-Based Engagement Navigator Service to Reduce CSC Disengagement
Brief Title: Hub-Based Engagement Navigator Service to Reduce CSC Disengagement
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Melanie E Bennett, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 1P01MH139228 (NIH)
Record Dates: First submitted 2024-09-01; First posted 2024-09-03 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Disengagement
Keywords: first episode psychosis; Coordinated Specialty Care; treatment disengagement; mental health services

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Engagement Navigator Service (ENS) (Experimental): ENS will be a centralized service, staffed by dedicated professional to (1) receive and organize referrals, (2) complete ongoing specialized training in engagement science and evidence-based strategies, (3) provide unbiased support when participants' and/or families' relationships with a CSC program are poor, (4) re-engage participants in CSC or actively connect them with other services if preferred, and (5) continue contact with those who refuse treatment in case they reconsider.
  Interventions: Other: Engagement Navigator Service (ENS)
- No ENS (No Intervention): Those who do not participate in ENS will comprise the no intervention arm.

INTERVENTIONS:
Other: Engagement Navigator Service (ENS) — ENS will be a centralized service, staffed by dedicated professional to (1) receive and organize referrals, (2) complete ongoing specialized training in engagement science and evidence-based strategies, (3) provide unbiased support when participants' and/or families' relationships with a CSC program are poor, (4) re-engage participants in CSC or actively connect them with other services if preferred, and (5) continue contact with those who refuse treatment in case they reconsider.
  Arms: Engagement Navigator Service (ENS)

SUMMARY:
This project will develop a hub-based engagement navigator service for participants and families at high risk for disengagement. The investigators will use robust Participatory Research methods to ensure integration of Coordinated Specialty Care (CSC) program staff, participants, and family members in developing all aspects of and materials for the service, conduct feasibility/acceptability testing in three CSC programs, and use this information to guide refinements. This will be followed by a mixed methods hub wide evaluation using a hybrid type I open cohort stepped wedge design to examine feasibility, acceptability, and effectiveness to improve disengagement outcomes and address target mechanisms.

DETAILED DESCRIPTION:
Coordinated Specialty Care (CSC) disengagement is alarmingly common and compromises the vision of CSC to support recovery in first episode psychosis (FEP; see Overall Section). The Early Psychosis Intervention Network's (EPINET) hub-based structure offers an opportunity to circumvent program-level implementation barriers by developing and implementing systems-level strategies to address disengagement. One strategy employs a centralized service, staffed by dedicated professionals working across a hub, to (1) receive and organize referrals, (2) complete ongoing specialized training in engagement science and evidence-based strategies, (3) provide unbiased support when participants' and/or families' relationships with a CSC program are poor, (4) re-engage participants in CSC or actively connect them with other services if preferred, and (5) continue contact with those who refuse treatment in case they reconsider. Currently, no hub-based strategy exists to address disengagement. The primary objective of this project is to use participatory research methods within a learning health system research framework to develop and evaluate a hub-based Engagement Navigator Service (ENS) to prevent CSC disengagement. The central hypothesis is that, once developed, ENS will support more months in treatment and lower disengagement rates than usual care (UC). The long-term goal is to co-produce a hub-based navigator service to reduce disengagement. The investigators will attain these objectives via the following specific aims:

Specific Aim 1. To develop ENS in partnership with the AC's Lived Experience and Family Member Collectives and CSC Program Implementation Subunit. Using participatory research, the investigators will specify ENS structure, training, and procedures for referrals. This aim will create the tools and resources needed to implement ENS at the hub-level.

Specific Aim 2. To conduct mixed methods feasibility/acceptability testing in three CSC programs. The investigators will track rates of and reasons for referral, length of time for navigators to contact and engage participants, and track needs that navigators address. The investigators will collect participant input via qualitative interviews. In this aim, feasibility and acceptability data and intervention experiences will be used to refine ENS.

Specific Aim 3. To conduct a mixed methods evaluation of ENS offered hub wide. Specific Aim 3a. In a hybrid type I, stepped wedge cluster randomized controlled trial, determine if access to ENS decreases disengagement compared to UC and improves target mechanisms. H1: Time in treatment for CSC participants with ENS access will be significantly longer than in UC. H2: Rate of disengagement for CSC participants with ENS access will be significantly lower than in UC. H3: Measures of autonomy, competence, and relatedness will be significantly higher for CSC participants with ENS access compared to UC. H4 (Exploratory): Autonomy, competence, and relatedness scores will mediate the treatment effect. Specific Aim 3b. Using a multi-stakeholder mixed methods process evaluation, examine feasibility, fidelity, and acceptability of ENS and identify implementation barriers and facilitators. This aim will evaluate ENS and detail experiences offering it across CLHS. This will prepare us to conduct a larger trial in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving services at Coordinated Specialty Care programs for the treatment of early episode psychosis
* Age 13-35

Exclusion Criteria:

* Do not meet inclusion criteria

Ages: 13 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 555 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Rate of discharge | From enrollment to end of treatment at 2 years
  The investigators will compare rate of disengagement for CSC participants with ENS access to those in usual care who do not have ENS access.
Time in treatment | From enrollment to end of treatment at 2 years
  The investigators will compare time in treatment for participants with ENS access to that of participants in usual care who do not have ENS access.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No